CLINICAL TRIAL: NCT02131194
Title: The Post-Vitrectomy Lenstatin Study: A Prospective Randomized Double Blind Human Clinical Trial Testing the Efficacy of Lenstatin in Inhibiting Cataract Formation and Progression After Pars Plana Vitrectomy
Brief Title: The Post-Vitrectomy Lenstatin™ Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lenstatin LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1-tunis
Record Dates: First submitted 2014-05-02; First posted 2014-05-06 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-12

CONDITIONS: Cataract, Nuclear Progressive
Keywords: Cataract; Nutritional Supplement
MeSH Terms: conditions — Cataract, Nuclear Progressive; Cataract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lenstatin (Experimental): Lenstatin (2) capsules orally per day for (6) months
  Interventions: Dietary Supplement: Lenstatin
- Sugar Pill (Placebo Comparator): Placebo manufactured to mimic Lenstatin (2) capsules orally per day for (6) months
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Lenstatin — Dietary Supplement Lenstatin
  Arms: Lenstatin
Drug: Placebo — Placebo sugar pill manufactured to mimic Lenstatin
  Arms: Sugar Pill

SUMMARY:
To determine the efficacy of Lenstatin™, an over-the-counter nutritional supplement, in inhibiting the progression of nuclear cataract in eyes after pars plana vitrectomy.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE

There are conflicting reports on the effectiveness of nutritional antioxidants in preventing or slowing the growth of age related cataracts, despite extensive laboratory evidence suggesting that oxidative damage to lens epithelial cells is a common underlying etiologic factor in cataractogenesis. One reported review of nine clinical trials involving over 117,000 patients suggested that beta-carotene, Vitamin E, and Vitamin C had no effect in preventing or slowing the progression of age-related cataract. Conversely, a randomized trial of over 14,000 US male physicians indicated that long-term daily multivitamin use modestly and significantly decreased the risk of cataract.

Cataract formation following pars plana vitrectomy is a well recognized post-operative complication of the procedure, with the reported incidence of clinically significant cataract development as high as 80% within 2 years after pars plana vitrectomy.

INVESTIGATIONAL AGENT

Lenstatin™ is a proprietary formulated nutritional supplement containing 11 micronutrients and anti-oxidants intended to be taken for the nutritional support of the human crystalline lens.

INTERVENTION

Participants will be randomized to treatment with Lenstatin or Placebo for (6) months following pars plana vitrectomy.

STUDY METHODS

Participants will have baseline nuclear density (cataract) measurements using the Pentacam Nucleus Staging (PNS) program. The Pentacam Scheimpflug imaging system is a non-contact and non-invasive anterior segment imaging device which has been shown to provide an immediate, quantitative, examiner-independent measurement of lens density which correlates with the LOCS III cataract grade. Serial Pentacam nuclear density measurements will be taken on each participant at (1) month intervals for (6) months.

ELIGIBILITY:
Inclusion Criteria:

* Adults over the age of 18
* Post pars plana vitrectomy surgery

Exclusion Criteria:

* Pediatric patients under the age of 18
* Pregnant women
* Hypersensitivity to any of the ingredients in Lenstatin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Pentacam Nuclear Density Measurements | (6) months
  The endpoint for determining the efficacy of Lenstatin in inhibiting cataract growth is a 95% confidence level of a statistically significant greater than 5% reduction in the rate of of increase in Pentacam nuclear density measurements in the Lenstatin™ treatment group compared to the placebo treatment group at 6 months postoperative pars plana vitrectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Scott W Tunis, MD FACS, Principal Investigator — Lenstatin LLC
Locations (1):
- Scott W. Tunis MD FACS, Wilmington, North Carolina, United States